CLINICAL TRIAL: NCT00867893
Title: d Immobilization Test (SIT) Test for Early Detection of Restless Legs Syndrome (RLS) Augmentation - Proof of Concept
Brief Title: Suggested Immobilization Test (SIT) Test for Early Detection of Restless Legs Syndrome (RLS) Augmentation - Proof of Concept
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Richard Allen, Research Associate, Department of Neurology, Johns Hopkins University
Other Study IDs: Sit-AUG
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- DA group: RLS patients started treatment on dopamine agonists within the past year
- NonDA: RLS patients started treatment on medication other than dopamine agonists within the past year

SUMMARY:
Some medications used to treat the restless legs syndrome (RLS) when taken for some time make the condition worse. This study seeks to find a method for early detection of this problem so that it can either be prevented or corrected.

DETAILED DESCRIPTION:
Long term dopaminergic treatment of RLS produces an exacerbation of RLS symptoms worse than before treatment for a significant percentage (5 - 70%) of those treated. This appears to be related to half-life, dose and duration of treatment. Shorter half-life medications appear to produce more augmentation. Once started augmentation appears to be progressive in many of the patients with the end result that the patient has much more severe RLS symptoms than before treatment. These symptoms can still be temporarily reduced by adding more dopaminergic treatment, but eventually this fails to suffice even with very high dopaminergic doses. The problem is finding a way to detect augmentation early during dopamine treatment both to determine the true rate of occurrence of this problem and to change treatment strategies before the problem becomes severe.

The suggested immobilization test creates the stimulus situation of protracted rest while lying down that provokes RLS symptoms. It provides a sensitive test for the severity of the symptom.. It should therefore provide an early detection of any exacerbation of symptoms such as that occurring with RLS augmentation.

In addition diphenhydramine also creates an exacerbation of RLS symptoms. This exacerbation would amplify the current severity of the RLS and as such could provide a tool for enhancing the degree of augmentation. Thus testing with a diphenhydramine challenge dose before the SIT test could provide an even more sensitive measure of augmentation

The investigators specifically hypothesize:

1. The objective measures from the SIT test will reveal an increase in severity of RLS that occurs with RLS augmentation at the same time or before the augmentation is detected by the usual subjective clinical assessments.
2. An oral dose of 25 mg of diphenhydramine taken 45 minutes before a SIT test will amplify the augmentation effects shown on the objective measures of the SIT. This will provide an enhanced detection of augmentation before or at the same time as that detected by either the SIT test alone or the clinical evaluation.

This study may for the first time provide a standard highly repeatable objective measure of RLS augmentation that is as or more sensitive as a very careful clinical evaluation by someone well trained in detecting RLS augmentation. As such it would prove clinically useful to evaluate RLS treatment progress. It would also provide an efficient method for evaluating the augmentation potential of new medications for RLS. .

ELIGIBILITY:
Inclusion Criteria:

1. Primary RLS (exclude all secondary RLS including those related to neuropathies and medications)
2. Adult and adolescents 18 years of age or older
3. One of the following 2 criteria must be met:

   * RLS treatment with either ropinirole or pramipexole or with a non-DA treatment (opioid or GABA active hypnotic), with the first dose each day taken at or before 4:30 PM. (Note this allows patients to be entered who had the usual tapered withdrawal from another medication with a concurrent gradual start of the DA agonist or opioid over a period of up to 12 months. In all such cases the initial evaluations must occur at least 6 weeks after discontinuing any prior drug treatment.) OR
   * Off all RLS medication treatments for at least 6 weeks AND planning on starting DA agonist or a non-DA treatment (opioid or GABA active hypnotic) as the only RLS medication treatment.

Exclusion Criteria:

1. Pregnant or lactating.
2. Inadequate birth control if female and able to become pregnant.
3. History of allergic reaction to diphenhydramine.
4. History of major psychiatric or chronic neurological disorder that would affect RLS treatment or judgment. These include but are not limited to bipolar depression, major affective disorder, schizophrenia, obsessive-compulsive disorder, and all neurodegenerative diseases.
5. History of another major sleep disorder other than RLS and insomnia: narcolepsy, significant sleep-disordered breathing (DBR>15/hr), and circadian rhythm disorder.
6. History of use of dopamine antagonist within the last year for any reason other than treating nausea.
7. History of use of tramadol within the last 3 months.
8. Unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RLS patients treated with medication
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2009-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Periodic Leg Movement/Hour on SIT PSG | 1 Month
  Occurs one month after Baseline SIT.
Periodic Leg Movement/Hour on SIT PSG | 2 Month
  Occurs 2 months after Baseline SIT.
Periodic Leg Movement/Hour on SIT PSG | 4 Month
  Occurs 4 months after Baseline SIT.
Periodic Leg Movement/Hour on SIT PSG | Month 6
  Occurs 6 months after Baseline SIT.
Periodic Leg Movement/Hour on SIT PSG | Month 9
  Occurs 9 months after Baseline SIT.
Periodic Leg Movement/Hour on SIT PSG | 12 Month
  Occurs 12 months after Baseline SIT.
Periodic Leg Movement/Hour on SIT PSG | 0 months/Baseline
  First SIT used as a baseline, 1 or 2 days depending on participant's past experience with the test.

CONTACTS AND LOCATIONS:
Overall Officials: Richard P Allen, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States